CLINICAL TRIAL: NCT02054949
Title: Pilot Study of N-acetyl Cysteine for Refractory Generalized Epilepsy in Children With Autism
Brief Title: Treatment Resistant Epilepsy and N-Acetyl Cysteine
Acronym: TRE-NAC
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no eligible subjects located
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Barbara Gracious, Principal Investigator, Nationwide Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB12-00325
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-10

CONDITIONS: Autistic Disorder; Seizures; Irritability
Keywords: N-acetyl cysteine; Refractory Seizures
MeSH Terms: conditions — Autistic Disorder; Seizures | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N-Acetyl Cysteine (NAC) (Experimental): NAC will be started at 500 mg by mouth twice daily for the first 2 weeks, then increased to 500 mg in the am and 1000 mg in the pm for week 3, and then increased to 1000 mg am and pm for weeks 4 through 8. Subjects will be maintained at the highest tolerated dose.
  Interventions: Drug: N-Acetyl Cysteine (NAC)

INTERVENTIONS:
Drug: N-Acetyl Cysteine (NAC) — NAC will be started at 500 mg by mouth twice daily for the first 2 weeks, then increased to 500 mg in the am and 1000 mg in the pm for week 3, and then increased to 1000 mg am and pm for weeks 4 through 8. Subjects will be maintained at the highest tolerated dose.

SUMMARY:
This is a study to find out whether the dietary amino acid supplement, N-acetyl cysteine (NAC) is helpful in reducing the frequency of seizures in children with autism and comorbid epilepsy whose seizures are not responding well to usual medical treatment. The study is also looking to see if this supplement is helpful for immediate and ongoing treatment of symptoms of irritability. Additionally, this study will also look to see if certain substances in the blood that measure a specific type of stress on cells in the body can help tell us how NAC may be helping.

DETAILED DESCRIPTION:
One third of patients with idiopathic autism have treatment resistant epilepsy, associated with earlier onset of seizures. In addition to insufficient response to medical treatment, they also have poorer responses to surgical and VNS approaches (Sansa et al 2011). Novel approaches to reduce seizure burden and improve quality of life for the children and their caregivers are needed.

There is a plethora of basic research documenting elevated oxidative stress in animal models of seizures. Several animal models have decreased oxidative stress through using compounds with antioxidant effects, but suprisingly, few human studies have been done to date.

This small open-label pilot study will examine the use of N-acetyl cysteine, an inexpensive but readily available over-the-counter nutritional supplement, to reduce seizure frequency in 10 youth with autism who have not responded completely to conventional anticonvulsant therapy

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents/young adults ages 6-21, male or female, all races and ethnicities.
2. Autism
3. IQ less than 80
4. 10 subjects with treatment resistant generalized epilepsy as defined by trials of 3 or more anticonvulsants with continued seizure frequency of at least 1 per week, need to use a helmet, or vagal nerve stimulator placement.
5. Children with at least 1 grand mal/generalized seizure per week.

Exclusion Criteria:

1. Inability to swallow capsules
2. In females, pregnancy or sexual activity
3. Daily acetaminophen, glucocorticoid, or nonsteroidal anti-inflammatory drugs, or daily NAC or high-dose antioxidant vitamin supplements within 30 days of baseline.
4. History of acute or chronic liver, renal, endocrine, infectious, autoimmune, hematologic, metabolic, or other disorder in the judgement of the study physician.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 year
  screening to enrollment and retention rates will be measured

SECONDARY OUTCOMES:
seizure frequency | up to 8 weeks
  seizure count

OTHER OUTCOMES:
side effect rating form for children and adolescents | at baseline, 4, and 8 weeks
  parent and child will be queried about changes in physical and mental health between study visits using a standardized form.
Aberrant Behavior Checklist | baseline, 4, and 8 weeks
  58 item parent-completed questionnaire
Autism Spectrum Rating Scale | baseline, 4, and 8 weeks
  parent report form on symptoms and behaviors in autism
oxidative stress measures | baseline, 4, and 8 weeks
  blood is collected and analyzed for oxidative changes in lipids, proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Gracious, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States